CLINICAL TRIAL: NCT03226041
Title: The Application of Transcutaneous CO2 Partial Pressure Monitoring in the Anesthesia of Patients Undergoing Retroperitoneoscopic Urologic Surgery
Brief Title: PTCCO2 Monitoring During Retroperitoneoscopic Urologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-SR-108
Record Dates: First submitted 2017-07-02; First posted 2017-07-21 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Transcutaneous Carbon Dioxide Partial Pressure Monitoring; Retroperitoneoscopic Urologic Surgery
Keywords: transcutaneous carbon dioxide; retroperitoneoscopic; urologic surgery; anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- retroperitoneoscopic urologic surgery (Experimental): All included patients will undergo retroperitoneoscopic renal or adrenal surgery with the transcutaneous carbon dioxide monitor.
  Interventions: Device: transcutaneous monitor (TCM-4 monitor)

INTERVENTIONS:
Device: transcutaneous monitor (TCM-4 monitor) — TCM-4 monitor, which had changed new electrode membrane and was calibrated by the same person(who had been trained systematically) before each placement. The electrode should be heated to 44℃, then fixed it to the anterior part of chest in the location of lateral position after remove grease by alcohol. The positon of electrode must be changed every 2 hours in order to avoid thermal injury, and should be calibrated again.

SUMMARY:
To investigate the accuracy and correlation of estimating arterial CO2 pressure（PaCO2） using a transcutaneous CO2 pressure（PTCCO2） monitor in patients undergoing retroperitoneoscopic renal or adrenal surgery.

DETAILED DESCRIPTION:
30 patients undergoing retroperitoneoscopic renal or adrenal surgery were included in this study.Their PaCO2, PetCO2, and PTCCO2values were measured at 3 time points before and 30min, 60min after pneumoperitoneum and calculated the different between each measure(PetCO2 and PTCCO2) and PaCO2. Agreement among measures was assessed by the Bland-Altman method.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing retroperitoneoscopic renal or adrenal surgery
2. Age more than 16 years.

Exclusion Criteria:

1. Care taker unable or unwilling to give oral informed consent
2. Patients with history of severe trauma, operations, smoking, and severe cardiovascular or respiratory diseases, such as coronary heart disease, congestive heart failure, or chronic obstructive pulmonary disease

4.Subject has a condition or allergy which would prohibit placing the probe 5.Subject has participated in a trial with any experimental drug or device trial within 30 days prior to enrollment in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Bias and precision of the transcutaneous carbon dioxide measurements | 0 minutes(baseline)
  correlation and agreement between PetCO2 and PaCO2 and PTCCO2
Bias and precision of the transcutaneous carbon dioxide measurements | 30 minutes
  correlation and agreement between PetCO2 and PaCO2 and PTCCO2
Bias and precision of the transcutaneous carbon dioxide measurements | 60 minutes
  correlation and agreement between PetCO2 and PaCO2 and PTCCO2

SECONDARY OUTCOMES:
complication: appearance of signs of thermal injury (redness, skin erythema, blisters, necrosis) under application of transcutaneous sensor temperatures of 44°C ) | 0 minutes(baseline)
  While the sensor temperatures heated to 44°C, the skin will be closely observed for any kind of thermic tissue damage
complication: appearance of signs of thermal injury (redness, skin erythema, blisters, necrosis) under application of transcutaneous sensor temperatures of 44°C ) | 30 minutes
  While the sensor temperatures heated to 44°C, the skin will be closely observed for any kind of thermic tissue damage
complication: appearance of signs of thermal injury (redness, skin erythema, blisters, necrosis) under application of transcutaneous sensor temperatures of 44°C ) | 60 minutes
  While the sensor temperatures heated to 44°C, the skin will be closely observed for any kind of thermic tissue damage

CONTACTS AND LOCATIONS:
Overall Officials: Shijiang Liu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided